CLINICAL TRIAL: NCT02513563
Title: A Phase II Trial of AZD1775 Plus Carboplatin-Paclitaxel in Squamous Cell Lung Cancer
Brief Title: AZD1775 Plus Carboplatin-Paclitaxel in Squamous Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18304
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Results first posted 2024-01-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: Squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Paclitaxel; adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carboplatin/Paclitaxel/AZD1775 (Experimental): Treatment: Combination of AZD1775 plus carboplatin and paclitaxel. Participants will be treated with this combination of drugs twice daily on days 1 and 2 and once on day 3 for a total of 5 doses during each 21 day cycle of treatment.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: AZD1775

INTERVENTIONS:
Drug: Carboplatin — Participants will be treated with carboplatin (area under the curve 5 (AUC5) will be used to determine the dosage) twice daily, days 1 and 2 and once a day on day 3 (5 doses) during each 21 day cycle of treatment.
  Other Names: Paraplatin®
Drug: Paclitaxel — Participants will be treated with paclitaxel 175 mg/m^2 twice daily, days 1 and 2 and once a day on day 3 (5 doses) during each 21 day cycle of treatment.
  Other Names: TAXOL®
Drug: AZD1775 — Participants will receive AZD1775 225 mg twice daily, days 1 and 2 and once a day on day 3 (5 doses) during each 21 day cycle of treatment.
  Other Names: MK1775

SUMMARY:
The purpose of this study is to find out what effects (good and bad) AZD1775 used in combination with carboplatin and paclitaxel will have on participants and their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Histologic or cytological diagnosis of Squamous Cell Lung Cancer (SQCLC) with advanced/metastatic stage, with no known curative treatment options. Prior platinum-containing adjuvant, neoadjuvant, or definitive chemoradiation therapy given for locally advanced disease is considered first line therapy only if recurrent (local or metastatic) disease developed within 6 months of completing therapy. Potential participants with recurrent disease > 6 months will be eligible.
* Female or male aged >/= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0/1
* Prior chemotherapy in the adjuvant setting is allowed
* Prior radiotherapy is allowed
* Any prior palliative radiation must have been completed at least 7 days prior to the start of the studies drugs and participants must have been recovered from any acute adverse effects prior to the start of the study treatment
* Prior Immunotherapy with PD1i, PDL1i, anti-CTLA -4 or vaccines is allowed
* Must have normal organ and marrow function
* Have archival tissue available or undergo a fresh biopsy where clinically feasible after discussion with the sponsor
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation and women who are breast feeding are excluded from the study. Both women and men should be fully informed of the lack of reproductive toxicity testing, and women must have a negative pregnancy test prior to enrollment.

Exclusion Criteria:

* Progressive, symptomatic untreated brain metastases
* Pregnancy or breast feeding
* A serious uncontrolled medical disorder or active infection that in the investigator's opinion would impair the participant's ability to receive study treatment
* Prior use of platinum or paclitaxel for stage IV Non-small Cell Lung Cancer (NSCLC) or concurrent use of other anticancer approved or investigational agents
* Use of anti-cancer treatment drug ?21 days or 5 half-lives (whichever is shorter) prior to the first dose of AZD1775. For drugs for which 5 half-lives is <21 days, a minimum of 10 days between termination of the prior treatment and administration of AZD1775 treatment is required.
* Major surgical procedures ?28 days of beginning study treatment, or minor surgical procedures ?7 days. No waiting period required following port-a-cath or other central venous access placement.
* Grade >1 toxicity from prior therapy EXCEPT: Alopecia, anorexia, and/or endocrinopathies on replacement therapy.
* Unable to swallow oral medications. Note: Patient may not have a percutaneous endoscopic gastrostomy (PEG) tube or be receiving total parenteral nutrition (TPN).
* Known Hepatitis B or C or HIV infection
* Second primary malignancy, other than in situ malignancies or adequately treated basal cell carcinoma of the skin or other malignancy treated at least 2 years previously with no evidence of recurrence
* Any of the following cardiac diseases currently or within the last 6 months: unstable angina pectoris, acute myocardial infarction, congestive heart failure > Class 2 (as defined by New York Heart Association (NYHA)), conduction abnormality not controlled with pacemaker or medication, significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
* Have had prescription or non-prescription drugs or other products (i.e., grapefruit juice) known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors or inducers of CYP3A4, which cannot be discontinued 2 weeks before Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug
* Co-administration of aprepitant and fosaprepitant during this study is prohibited
* AZD1775 is an inhibitor of breast cancer resistance protein (BCRP). The use of statins including Atorvastatin which are substrates for BCRP are therefore prohibited and patients should be moved on to non-BCRP alternatives
* Herbal preparations are not allowed throughout the study. These herbal medications include, but are not limited to: St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng
* History of Torsades de pointes unless all risk factors that contributed to Torsades have been corrected
* Mean resting corrected QTc interval using the Fridericia formula (QTcF) >450 msec/male and >470 msec/female (as calculated per institutional standards) obtained from 1 electrocardiograms (ECGs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle Gray, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboplatin/Paclitaxel/AZD1775
Started | 42
Completed | 33
Not Completed | 9
Not completed — Death | 4
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin/Paclitaxel/AZD1775
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 40
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is measured from date of first study treatment to death, progression of disease, or the last follow-up data, whichever comes first. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 2 years
Population: Evaluable participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel/AZD1775
Number analyzed (Participants) | 41
months | 4.8 [4.1 to 5.7]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration of time from the date for first treatment (Cycle 1 Day 1) to the date of death.
Time Frame: Up to 2 years
Population: Evaluable participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel/AZD1775
Number analyzed (Participants) | 41
months | 7.3 [6.4 to 8.4]

3. Secondary Outcome: Duration of Overall Response (OR)
Description: The duration of overall response is measured from the time measurement criteria are met for Complete Response (CR) or Partial Response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 2 years
Population: Evaluable participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel/AZD1775
Number analyzed (Participants) | 14
months | 4.4 [3.2 to 4.9]

4. Secondary Outcome: Percentage of Participants With Disease Control
Description: DCR: Complete Response (CR), Partial Response (PR), and Stable Disease (SD).
Time Frame: Up to 2 years
Population: Evaluable participants
Measure: Number (80% Confidence Interval); unit: percentage
Arm/Group | Carboplatin/Paclitaxel/AZD1775
Number analyzed (Participants) | 41
percentage | 61 [51 to 71]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were collected from date of consent until 4 weeks after last study treatment. Adverse Events were collected from treatment Cycle 1 day 1 until 4 weeks after last study treatment. Events were collected an average of 129 days.
Arm/Group | Carboplatin/Paclitaxel/AZD1775
All-Cause Mortality (participants affected / at risk) | 4/42
Serious Adverse Events (participants affected / at risk) | 26/42
Other Adverse Events (participants affected / at risk) | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel/AZD1775 (N=42)
Lung infection (Infections and infestations) | 5 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions -Other (General disorders) | 1 (1) — Pain from left gluteal mass
Generalized edema (General disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Death NOS (General disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Seizure (Nervous system disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 1 (1) — Salmonella
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Heart failure (Cardiac disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Pancytopenia (Investigations) | 2 (2)
Pleural infection (Infections and infestations) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Chest pain - Cardiac (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders -Other (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pericardial tamponade (Cardiac disorders) | 1 (1)
Pain in extremity (General disorders) | 1 (1) — bilateral lower extremity pain due to venous thrombosis
Esophagitis (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel/AZD1775 (N=42)
Diarrhea (Gastrointestinal disorders) | 21 (34)
Nausea (Gastrointestinal disorders) | 20 (31)
Vomiting (Gastrointestinal disorders) | 12 (16)
Abdominal Pain (Gastrointestinal disorders) | 9 (10)
Constipation (Gastrointestinal disorders) | 7 (8)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 21 (37)
Pain (General disorders) | 10 (14)
Infusion related reaction (General disorders) | 6 (9)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (9)
Hyponatremia (Metabolism and nutrition disorders) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 17 (28)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 7 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (4)
Dizziness (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 2 (2)
Aphonia (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (5)
Investigations - Other (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 2 (4)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (4)
Weight loss (Investigations) | 1 (2)
Infections and infestations - Other (Infections and infestations) | 3 (4)
Lung infection (Infections and infestations) | 3 (6)
Upper respiratory infection (Infections and infestations) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Cardiac disorders - Other (Cardiac disorders) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (3)
Confusion (Psychiatric disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT02513563/Prot_SAP_000.pdf